CLINICAL TRIAL: NCT02961348
Title: Timing of Oral Anticoagulant Therapy in Acute Ischemic Stroke With Atrial Fibrillation: a Prospective Multicenter Registry-based Non-inferiority Randomized Controlled Clinical Trial
Brief Title: TIMING of Oral Anticoagulant Therapy in Acute Ischemic Stroke With Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: The Swedish Stroke Register (Riksstroke) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: U-2015-341; 2015-00881 (Other Grant/Funding Number: The Swedish Research Council)
Record Dates: First submitted 2016-11-08; First posted 2016-11-10 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Ischemic Stroke; Atrial Fibrillation
Keywords: Oral anticoagulants (NOAC)
MeSH Terms: conditions — Ischemic Stroke; Atrial Fibrillation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early start of NOAC (Active Comparator): Day 1 to day 4 after ischemic stroke onset
  Interventions: Other: Early start of NOAC
- Late start of NOAC (Active Comparator): Day 5 to day 10 after ischemic stroke onset
  Interventions: Other: Late start of NOAC

INTERVENTIONS:
Other: Early start of NOAC — Initiation of NOAC up until day 4 after acute ischemic stroke in patients with atrial fibrillation
  Arms: Early start of NOAC
Other: Late start of NOAC — Initiation of NOAC between day 5 and day 10 after acute ischemic stroke in patients with atrial fibrillation
  Arms: Late start of NOAC

SUMMARY:
This study will compare early with late start of treatment with Non-vitamin K oral anticoagulation (NOAC) in adult patients with acute ischemic stroke and atrial fibrillation; it is a registry-based randomized clinical trial (R-RCT) using The Swedish Stroke Register (Riksstroke). Half of the patients will start NOAC early (within 4 days after stroke onset) while the other half will start late (5-10 days after stroke onset).

DETAILED DESCRIPTION:
Oral anticoagulation therapy is well established and highly recommended for the prevention of recurrent ischemic stroke in patients with atrial fibrillation, but the optimal time point to start after an acute ischemic stroke is not known.

The intervention in this study will be timing of treatment onset. The choice of NOAC (i.e. apixaban, dabigatran, edoxaban or rivaroxaban) after the acute ischemic stroke is at the discretion of the treating physician.

This study will use the Swedish Stroke Register for enrolment, randomization and follow-up, with additional data linkage from other mandatory national registers. Primary outcome will be assessed at 90 days and secondary outcomes (including all-cause mortality and health economic analyses) and will be assessed at 90 days and up to one year after the index ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years) with acute ischemic stroke and atrial fibrillation
* Eligible and willing to start (or re-start) NOAC
* Registered in The Swedish Stroke Register
* Signed informed consent

Exclusion Criteria:

* Contraindication to NOAC (e.g. ongoing bleeding, mechanical heart valve prosthesis)
* Ongoing therapy with NOAC (without ≥2 days interruption at index stroke)
* International normalized ratio (INR)>1.7
* No second brain imaging (CT/MRI) after thrombolysis/thrombectomy
* Previous randomization in the TIMING study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 888 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Composite outcome of recurrent ischemic stroke, symptomatic intracerebral hemorrhage, or all-cause mortality | 90 days

SECONDARY OUTCOMES:
Recurrent acute ischemic stroke | 90 days
  Defined as a new focal neurological deficit of sudden onset lasting at least 24 h (or <24 h if following therapeutic intervention, i.e. thrombolysis or thrombectomy, or if the deficit results in death < 24 h), occurring >24 hours after the index ischemic stroke, irrespective of vascular territory and that is not attributable to edema, brain shift, hemorrhagic transformation, intercurrent illness, hypoxia, or drug toxicity
Symptomatic intracerebral hemorrhage (S-ICH) | 90 days
  Defined as a new focal neurological deficit of sudden onset lasting at least 24 h with documented intracerebral hemorrhage (ICH) on imaging (computed tomography (CT) or magnetic resonance imaging (MRI)). Any intraparenchymal hematoma (≥10mm) will be considered, including hemorrhagic transformation of the index ischemic stroke. However microhemorrhages (<10mm) are not considered to be an ICH. ICH will be classified as symptomatic if it is associated with ≥4 points in total NIHSS or ≥2 points in one NIHSS category
All-cause mortality | 90 days
Functional outcome | 90 days
  Defined by grade on the modified Rankin Scale (mRS)
Major hemorrhages | 90 days
  Defined as bleedings that are fatal or life-threatening (according to the definition by the International Society on Thrombosis and Haemostasis) or lead to hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Oldgren, MD. PhD, Principal Investigator — Dept of Medical Sciences, Uppsala University, Sweden; Signild Åsberg, MD. PhD, Principal Investigator — Dept of Medical Sciences, Uppsala University, Sweden
Locations (36):
- Sweden (36):
  - Alingås Hospital, Alingsås
  - Enköping Hospital, Enköping
  - Mälarsjukhuset Hospital, Eskilstuna
  - Falu Hospital, Falun
  - Gävle Hospital, Gävle
  - Sahlgrenska University Hospital Östra, Gothenburg
  - Sahlgrenska University Hospital, Gothenburg
  - Hallands Hospital, Halmstad
  - Hässleholm Hospital, Hässleholm
  - Helsingborg Hospital, Helsingborg
  - Karolinska University Hospital - Huddinge, Huddinge
  - Hudiksvalls sjukhus, Hudiksvall
  - Ryhov, Jönköping
  - Kalmar Hopsital, Kalmar
  - Länssjukhuset Kalmar, Kalmar
  - Kiruna Hospital, Kiruna
  - Köping Hospital, Köping
  - Kungälv Hospital, Kungälv
  - Lindesberg Hospital, Lindesberg
  - Lund, Lund
  - Malmö University Hospital, Malmo
  - Motala Hospital, Motala
  - Sahlgrenska Universitetssjukhuset Mölndal, Mölndal
  - Nyköping Hospital, Nyköping
  - Oskarshamn Hospital, Oskarshamn
  - Örebro University Hospital, Örebro
  - Skaraborg Hospital, Skövde
  - Karolinska University Hospital, Solna
  - Capio S:t Görans Hospital, Stockholm
  - Danderyd University Hospital, Stockholm
  - Södersjukhuset, Stockholm
  - Sundsvall County Hospital, Sundsvall
  - University Hospital of Umeå, Umeå
  - Uppsala University Hospital, Uppsala
  - Hallands Hospital, Varberg
  - Västerås Hospital, Västerås

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Asberg S, Hijazi Z, Norrving B, Terent A, Ohagen P, Oldgren J. Timing of oral anticoagulant therapy in acute ischemic stroke with atrial fibrillation: study protocol for a registry-based randomised controlled trial. Trials. 2017 Dec 2;18(1):581. doi: 10.1186/s13063-017-2313-9. PMID 29197413
- [Result] Oldgren J, Asberg S, Hijazi Z, Wester P, Bertilsson M, Norrving B; National TIMING Collaborators. Early Versus Delayed Non-Vitamin K Antagonist Oral Anticoagulant Therapy After Acute Ischemic Stroke in Atrial Fibrillation (TIMING): A Registry-Based Randomized Controlled Noninferiority Study. Circulation. 2022 Oct 4;146(14):1056-1066. doi: 10.1161/CIRCULATIONAHA.122.060666. Epub 2022 Sep 6. PMID 36065821